CLINICAL TRIAL: NCT02241759
Title: A Phase I, Single-Centre, Randomised, Placebo and Positive- Controlled, Parallel-Group Study of the Electrocardiographic Effects of TA-8995 in Healthy Male and Female Subjects
Brief Title: Study of the Electrocardiographic Effects of TA-8995
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Xention Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TA-8995-04
Record Dates: First submitted 2014-08-20; First posted 2014-09-16 (Estimated); Last update posted 2015-02-16 (Estimated); Status verified 2015-02

CONDITIONS: Dyslipidaemia
MeSH Terms: conditions — Dyslipidemias | interventions — TA-8995; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- TA-8995 (Experimental): Single oral dose of 150mg TA-8995
  Interventions: Drug: TA-8995
- Placebo (Experimental): Single oral dose of placebo to TA-8995
  Interventions: Drug: Placebo
- Moxifloxacin (Active Comparator): Single open-label oral dose of 400mg moxifloxacin
  Interventions: Drug: Moxifloxacin

INTERVENTIONS:
Drug: TA-8995
  Arms: TA-8995
Drug: Moxifloxacin
  Arms: Moxifloxacin
Drug: Placebo
  Arms: Placebo

SUMMARY:
A study in healthy males and females to see if a high single dose of TA-8995 has an effect on the ECG QTcF interval.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or females of non-child bearing potential

Exclusion Criteria:

* Receiving any other drug therapy
* Clinically significant medical history
* Abnormal ECGs or vital signs

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 136 (Actual)
Dates: Start 2014-08; Primary Completion 2014-11 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline in QT interval corrected for heart rate (QTc) for TA-8995 versus placebo | 4 days

SECONDARY OUTCOMES:
Relationship between plasma levels of TA-8995 and the QTcF effect | 4 days

CONTACTS AND LOCATIONS:
Overall Officials: Ashley Brooks, Principal Investigator — Covance
Locations (1):
- Covance Clinical Research Unit Ltd, Leeds, United Kingdom